CLINICAL TRIAL: NCT01042743
Title: Laparoscopic Surgery Versus Robot Surgery for Right-side Colon Cancer: Short-term Outcome of a Randomised Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Colorectal Cancer Center, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNUHCRC001
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Colon Cancer
Keywords: colon cancer; robot; laparoscopy; primary, right-side colon cancer; robot-assisted surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAP (Experimental): individuals who underwent robot-assisted surgery for primary right-sied colon cancer
  Interventions: Procedure: robot-assisted surgery
- LAP (Active Comparator): Individuals who underwent laparoscopic surgery for primary right-side colon cancer
  Interventions: Procedure: laparoscopic right-hemicolectomy

INTERVENTIONS:
Procedure: robot-assisted surgery — da Vinci surgical system® (Intuitive Surgical, Sunnyvale, CA, USA)
  Arms: RAP
Procedure: laparoscopic right-hemicolectomy — Conventional laparoscopic procedures
  Arms: LAP

SUMMARY:
The recent introduction of robotic surgical system has revolutionized the field of minimally invasive surgery. The investigators hypothesized that adoption of a robotic surgical system for patients with right-side colon cancer seems appealing because This system provides high-definition three-dimensional vision, eliminates physiologic tremor, and better ergonomics. This randomized controlled trial was designed to determine the safety and efficacy of robotic right hemicolectomy in comparison with laparoscopic right hemicolectomy.

ELIGIBILITY:
Inclusion Criteria:

* primary cancer
* right-side located tumor (from cecum to proximal transverse colon)

Exclusion Criteria:

* tumor with obstruction
* tumor with perforation
* clinically advanced tumor (T4 stage)
* tumor with distant metastases
* synchronous tumor

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
surgical quality based on pathological examination | during perioperative period (1-30 days after operation)

SECONDARY OUTCOMES:
complication | during perioperative period ( 1-30 days after primary operation)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

REFERENCES:
- [Derived] Park JS, Lee SM, Choi GS, Park SY, Kim HJ, Song SH, Min BS, Kim NK, Kim SH, Lee KY. Comparison of Laparoscopic Versus Robot-Assisted Surgery for Rectal Cancers: The COLRAR Randomized Controlled Trial. Ann Surg. 2023 Jul 1;278(1):31-38. doi: 10.1097/SLA.0000000000005788. Epub 2023 Jan 3. PMID 36594748
- [Derived] Park JS, Choi GS, Park SY, Kim HJ, Ryuk JP. Randomized clinical trial of robot-assisted versus standard laparoscopic right colectomy. Br J Surg. 2012 Sep;99(9):1219-26. doi: 10.1002/bjs.8841. PMID 22864881